CLINICAL TRIAL: NCT00149500
Title: Social Support and Education in Asthma Follow-up (SSEA)
Acronym: SSEA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 259; R01HL072919 (NIH)
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Coaching group for lifestyle changes (Experimental): Patients received monthly phone calls with coaching for lifestyle changes over 2 years.
  Interventions: Behavioral: Coaching
- Routine pediatric care (No Intervention): This group receives routine care with their pediatrician.

INTERVENTIONS:
Behavioral: Coaching — Patients received monthly calls to assist in behavioral change relative to asthma care
  Arms: Coaching group for lifestyle changes

SUMMARY:
We will evaluate the effect of an eighteen-month asthma coaching intervention for parents/caregivers of children with asthma to reduce asthma morbidity. The primary objective is to determine if asthma coaching will significantly reduce asthma morbidity as measured by a reduction in the number of ED visits and hospitalizations for the children during the 18 months of active coaching and during the 18 months after the coaching stops.

We will provide half of the subjects (parents/caregivers) with access to assistance from an asthma coach for 18 months (including 2 contacts with an asthma nurse during the first 6 months). The other half of the subjects will not have an asthma coach, but their children will have their usual routine care with their primary care providers. The nurse and coach will help the subjects learn more about caring for their children's asthma and improving interactions with the primary care providers for their children.

DETAILED DESCRIPTION:
BACKGROUND:

Our previous NHLBI-supported study (HL 57232) showed that a combination treatment of "Coaching" through follow-up phone calls 2 and 5 days following an index ED visit plus monetary incentive was highly effective in increasing the percentage of low-income urban children who received recommended primary care within 2 weeks of the ED visit for asthma, 44% in the intervention group vs 29% in usual care (p = 0.0004). However, the intervention was not associated with significant differences in morbidity (subsequent ED visits). We conclude that the intervention was effective in promoting the initial link to primary care, but was not effective in sustaining that link or management practices to minimize acuity of symptoms during exacerbation.

DESIGN NARRATIVE:

Primary outcome The proportion of children of subjects in each group who have at least one ED visit for acute asthma symptoms during the thirty-six month period following enrollment.

Key secondary outcomes A. The proportion of children of subjects in each group who are hospitalized during the thirty-six month period following enrollment.

B. The proportion of children of subjects in each group who have either acute asthma visits or asthma-planning visits with their primary care providers.

C. The costs of asthma-related care during the thirty-six month period D. Variables which may mediate or moderate the intervention such as the attitudes toward asthma care of the subjects and the personal social support perceived by the subjects .

ELIGIBILITY:
Inclusion criteria:

A. The child of the parent/caregiver has a diagnosis of asthma made by a physician and reported by the parent, or diagnosis of asthma made during the ED visit if the child has experienced two previous wheezing episodes.

B. The child will undergo treatment during the enrollment ED visit for the current asthma exacerbation, as determined by the treating ED clinician. As a result, only parents/caregivers with children experiencing a significant wheezing episode will be entered into the study.

C. The child is 2-10 years of age (second birth date until, but not including, eleventh birth date).

D. The child has Medicaid or no medical insurance. This criterion permits easy identification and selection of low-income children/families, who are the target population for this proposal.

E. The parent/caregiver has a working telephone at home. F. The child attends one of the target practices (7 private practices and 5 federally funded clinics) for routine care.

G. The parent/caregiver and child live within the St. Louis metro area.

Exclusion criteria:

A. The child attends a practice other than the target group. B. The parent/caregiver and child live outside of the St. Louis metro area. C. The child has a chronic illness other than asthma that manifests as wheezing or respiratory symptoms.

D. The parent/caregiver does not have a working telephone in home. E. The parent/caregiver is not able to effectively communicate in English.

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 241 (Actual)
Dates: Start 2003-09; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
ER visits | 18 months
  Documenting the number of ER visits per patient in the 18 month period.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Strunk, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nelson KA, Highstein GR, Garbutt J, Trinkaus K, Fisher EB, Smith SR, Strunk RC. A randomized controlled trial of parental asthma coaching to improve outcomes among urban minority children. Arch Pediatr Adolesc Med. 2011 Jun;165(6):520-6. doi: 10.1001/archpediatrics.2011.57. PMID 21646584